CLINICAL TRIAL: NCT01667029
Title: A Single-center, Randomized, Double-blind Clinical Study to Evaluate the Effect of Sulfasalazine on Painful Neuropathy
Brief Title: Study of Sulfasalazine in Treating Painful Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brian Wainger, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-p-001443
Record Dates: First submitted 2012-08-14; First posted 2012-08-17 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-07

CONDITIONS: Painful Neuropathy
MeSH Terms: conditions — Neuropathy, Painful | interventions — Sulfasalazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sulfasalazine (Experimental): 1 g oral twice daily for 2 weeks
  Interventions: Drug: Sulfasalazine
- placebo (Placebo Comparator): oral placebo pill twice daily for two weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Sulfasalazine
  Arms: sulfasalazine
Drug: placebo
  Arms: placebo

SUMMARY:
The investigators hypothesize that sulfasalazine, an FDA-approved medication for rheumatoid arthritis and ulcerative colitis, may be beneficial in neuropathic pain conditions. In this study, the investigators will evaluate whether sulfasalazine improves pain due to painful peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Painful neuropathy
* Michigan Neuropathy Screening Instrument score of 3 or greater
* no obvious alternative explanation for neuropathy
* average baseline pain > 4/10

Exclusion Criteria:

* other severe pain
* anticipated difficulty weaning off medications
* past or current psychiatric disorder as determined by Mini International Neuropsychiatric Interview
* medical contraindication to sulfasalazine
* not proficient in English (due to heavy use of questionaires)
* pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Wainger, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sulfasalazine Then Placebo: Sulfasalazine (1 g oral twice daily) for two weeks, washout period of one week, placebo for 2 week period
- Placebo Then Sulfasalazine: Oral placebo pill twice daily for two weeks, washout period of one week, sulfasalazine for 2 week period
Period: Overall Study
Arm/Group | Sulfasalazine Then Placebo | Placebo Then Sulfasalazine
Started | 4 | 4
Completed | 3 | 3
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to either Group A or Group B:
  Group A: Placebo daily for two weeks, washout period of one week, sulfasalazine for 2 week period Group B: Sulfasalazine daily for two weeks, washout period of one week, placebo for 2 week period.
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (5.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Pain Score (First Treatment Period)
Description: Average pain score will be the average of daily pain scores (0-10) recorded by the subject in a pain diary during the second week of the two week treatment period. Higher scores are worse (0=no pain, 10=pain as bad as you can imagine).
Time Frame: second week of two week treatment period
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sulfasalazine: 1 g oral twice daily for 2 weeks
  Sulfasalazine
- Placebo: oral placebo pill twice daily for two weeks.
  placebo
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 4 | 4
units on a scale | 5.60 (1.35) | 4.20 (0.91)

2. Secondary Outcome: Pain Score (Using the Crossover Comparison Structure of the Study)
Description: as for outcome 1
Time Frame: Assessed at end of two week treatment period
Population: 8 participants were randomized, but 2 participants did not complete the second period of the study. So 6 participants received both sulfasalazine and placebo treatments, one only received sulfasalazine in period 1, and one only received placebo in period 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 7 | 7
units on a scale | 4.91 (1.38) | 3.93 (2.08)

3. Secondary Outcome: Number of Patients With >=50% Pain Reduction (First Treatment Period)
Description: Average pain score will be the average of daily pain scores (0-10) recorded by the subject in a pain diary at baseline and during the second week of the two week treatment period. Higher scores are worse (0=no pain, 10=pain as bad as you can imagine). Percent pain reduction will be calculated from BL to end of treatment period 1 (2 weeks), based on average pain scores at each time point.
Time Frame: second week of two week treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

4. Secondary Outcome: Number of Patients With >=50% Pain Reduction (Using the Crossover Comparison Structure of the Study)
Description: Average pain score will be the average of daily pain scores (0-10) recorded by the subject in a pain diary during baseline and the second week of each of the two week treatment periods. Higher scores are worse (0=no pain, 10=pain as bad as you can imagine). Percent pain reduction will be calculated from BL to end of treatment period 1 (2 weeks) and from end of treatment period 1 to end of treatment period 2 (2 weeks), based on average pain scores at each time point.
Time Frame: Assessed at end of two week treatment period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 7 | 7
Participants | 0 | 1

5. Secondary Outcome: Physical Functioning Score Assessed Using the Brief Pain Inventory (BPI) Interference Scale (First Treatment Period Only)
Description: The BPI interference items are general activity, mood, walking ability, normal work (including housework), relations with other people, sleep, and enjoyment of life. The seven items are rated from 0 (pain does not interfere) to 10 (pain completely interferes).
Time Frame: Assessed at end of two week treatment period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 4 | 4
units on a scale
  General activity | 5.25 (2.75) | 4.00 (1.41)
  Mood | 3.75 (3.86) | 5.00 (2.16)
  Walking ability | 4.50 (3.87) | 5.50 (2.08)
  Normal work | 5.25 (4.03) | 4.75 (2.50)
  Relations with other people | 1.25 (2.50) | 3.75 (1.71)
  Sleep | 5.00 (3.56) | 5.25 (2.22)
  Enjoyment of life | 5.75 (4.65) | 4.75 (2.50)

6. Secondary Outcome: Physical Functioning Score Assessed Using the Euroquality of Life (EQ-5D) Metrics (First Treatment Period Only)
Description: The EQ-5D physical functioning items are mobility self-care, and usual activities. These three items are rated from 1 (no problems) to 5 (unable).
Time Frame: Assessed at end of two week treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 4 | 4
Participants
  EQ-5D mobility: 1 | 1 | 1
  EQ-5D mobility: 2 | 1 | 2
  EQ-5D mobility: 3 | 2 | 0
  EQ-5D mobility: 4 | 0 | 1
  EQ-5D mobility: 5 | 0 | 0
  EQ-5D self-care: 1 | 3 | 4
  EQ-5D self-care: 2 | 1 | 0
  EQ-5D self-care: 3 | 0 | 0
  EQ-5D self-care: 4 | 0 | 0
  EQ-5D self-care: 5 | 0 | 0
  EQ-5D usual activities: 1 | 2 | 1
  EQ-5D usual activities: 2 | 1 | 1
  EQ-5D usual activities: 3 | 1 | 2
  EQ-5D usual activities: 4 | 0 | 0
  EQ-5D usual activities: 5 | 0 | 0

7. Secondary Outcome: Physical Functioning Score Assessed Using the Brief Pain Inventory (BPI) Interference Scale (Using the Crossover Comparison Structure of the Study)
Description: as for outcome 5
Time Frame: Assessed at end of two week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 7 | 7
units on a scale
  General activity | 4.00 (2.77) | 3.71 (2.06)
  Mood | 3.57 (3.10) | 4.00 (2.94)
  Walking ability | 3.57 (3.21) | 4.57 (2.57)
  Normal work | 4.14 (3.48) | 4.14 (2.61)
  Relations with other people | 1.43 (2.15) | 2.57 (1.99)
  Sleep | 4.86 (3.24) | 4.43 (2.76)
  Enjoyment of life | 4.57 (4.39) | 4.00 (3.61)

8. Secondary Outcome: Physical Functioning Score Assessed Using the Euroquality of Life (EQ-5D) (Using the Crossover Comparison Structure of the Study)
Description: as for outcome 6
Time Frame: Assessed at end of two week treatment period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 7 | 7
Participants
  EQ-5D mobility: 1 | 4 | 2
  EQ-5D mobility: 2 | 1 | 3
  EQ-5D mobility: 3 | 2 | 1
  EQ-5D mobility: 4 | 0 | 1
  EQ-5D mobility: 5 | 0 | 0
  EQ-5D self-care: 1 | 5 | 7
  EQ-5D self-care: 2 | 2 | 0
  EQ-5D self-care: 3 | 0 | 0
  EQ-5D self-care: 4 | 0 | 0
  EQ-5D self-care: 5 | 0 | 0
  EQ-5D usual activities: 1 | 4 | 2
  EQ-5D usual activities: 2 | 2 | 2
  EQ-5D usual activities: 3 | 1 | 3
  EQ-5D usual activities: 4 | 0 | 0
  EQ-5D usual activities: 5 | 0 | 0

9. Secondary Outcome: Emotional Functioning (First Treatment Period Only)
Description: Will be assessed by the Beck Depression Inventory (BDI) total score. The BDI has 21 items, each scored 0-3. Higher values are worse. The total score is the sum of the 21 items and ranges from 0-63.
Time Frame: Assessed at end of two week treatment period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 4 | 4
units on a scale | 8.25 (5.12) | 10.50 (6.61)

10. Secondary Outcome: Emotional Functioning (Using the Crossover Comparison Structure of the Study)
Description: as for outcome 9
Time Frame: Assessed at end of two week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 7 | 7
units on a scale | 7.29 (5.91) | 8.29 (6.29)

11. Secondary Outcome: Overall Improvement (First Treatment Period Only)
Description: The Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. Item 1 is as follows: Since beginning treatment at this clinic, how would you describe the change (if any) in ACTIVITY LIMITATIONS, SYMPTOMS, EMOTIONS, and OVERALL QUALITY OF LIFE, related to your painful condition? (tick ONE box) (1=No change (or condition has gotten worse), 2=Almost the same, hardly any change at all, 3=A little better, but no noticeable change, 4=Somewhat better, but the change has not made any real difference, 5=Moderately better, and a slight but noticeable change, 6=Better, and a definite improvement that has made a real and worthwhile difference, 7=A great deal better, and a considerable improvement that has made all the difference). Item 2 is as follows: In a similar way, please circle the number below that matches your degree of change since beginning care at this clinic (0-10 scale): 0= Much better, 5= No change, 10= Much worse.
Time Frame: Will be assessed at end of two week treatment period
Population: 2 participants in the sulfasalazine group are missing PGIC information.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 2 | 4
units on a scale
  PGIC Item 1 | 1.50 (0.71) | 1.75 (0.96)
  PGIC Item 2 | 5.00 (0.00) | 4.50 (1.00)

12. Secondary Outcome: Overall Improvement (Using the Crossover Comparison Structure of the Study)
Description: as for outcome 11
Time Frame: Will be assessed at end of two week treatment period
Population: 8 participants were randomized, but 2 participants did not complete the second period of the study. So 6 participants received both sulfasalazine and placebo treatments, one only received sulfasalazine in period 1, and one only received placebo in period 1. 2 of the sulfasalzine participants are missing PGIC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 5 | 7
units on a scale
  PGIC item 1 | 2.80 (2.39) | 3.00 (2.08)
  PGIC item 2 | 4.00 (1.73) | 3.56 (1.81)

13. Secondary Outcome: Categorical Rating of Pain Intensity (First Treatment Period Only)
Description: Assessed using number of days rated as none, mild, moderate, or severe in pain diary
Time Frame: Assessed at end of two week treatment period
Population: One participant in the sulfasalazine arm did not complete the categorical pain data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 3 | 4
days
  "None" rating | 0 (0) | 0 (0)
  "Mild" rating | 1.67 (2.89) | 1.75 (3.50)
  "Moderate" rating | 4.33 (2.52) | 5.25 (3.50)
  "Severe" rating | 1.00 (1.73) | 0 (0)

14. Secondary Outcome: Categorical Rating of Pain Intensity (Using the Crossover Comparison Structure of the Study)
Description: Assessed using number of days rated as none, mild, moderate, or severe in pain diary
Time Frame: Assessed at end of two week treatment period
Population: 8 participants were randomized, but 2 participants did not complete the second period of the study. So 6 participants received both sulfasalazine and placebo treatments, one only received sulfasalazine in period 1, and one only received placebo in period 1. One participant did not complete the categorical pain data in either period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 6 | 6
days
  "None" rating | 0 (0) | 1.17 (2.86)
  "Mild" rating | 2.00 (3.16) | 1.83 (2.99)
  "Moderate" rating | 4.33 (2.88) | 3.83 (3.54)
  "Severe" rating | 0.67 (1.21) | 0.17 (0.41)

15. Secondary Outcome: Breakthrough Treatment (First Treatment Period Only)
Description: Number of days breakthrough pain medication was taken
Time Frame: Assessed during two week treatment period
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 4 | 4
days | 0.75 (0.96) | 2.00 (2.83)

16. Secondary Outcome: Breakthrough Treatment (Using the Crossover Comparison Structure of the Study)
Description: Number of days breakthrough pain medication was taken
Time Frame: Assessed during two week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 7 | 7
days | 1.29 (2.21) | 1.14 (2.27)

17. Secondary Outcome: Missed Medication Dose (First Treatment Period Only)
Description: Number of missed medication doses
Time Frame: Assessed during two week treatment period
Measure: Mean (Standard Deviation); unit: dose
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 4 | 4
dose | 0 (0) | 0 (0)

18. Secondary Outcome: Missed Medication Doses (Using the Crossover Comparison Structure of the Study)
Description: Number of missed medication doses
Time Frame: Assessed during two week treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Sulfasalazine | Placebo
Number analyzed (Participants) | 7 | 7
doses | 0.43 (1.13) | 0 (0)

ADVERSE EVENTS:
Time Frame: Two study periods that were each two weeks in length.
Arm/Group | Sulfasalazine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulfasalazine (N=8) | Placebo (N=8)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT01667029/Prot_SAP_000.pdf